CLINICAL TRIAL: NCT02257463
Title: Effect of Inspiratory Muscle Training on Exercise Performance and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Dina Aboelkhair Abdallah, assistant lecturer in chest medicine, Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MD/4
Record Dates: First submitted 2014-09-26; First posted 2014-10-06 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; inspiratory muscle training; dyspnea; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Theophylline; Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Study group (group A) (Active Comparator): pharmacologic treatment: theophylline "uniphyllin", long acting bronchodilators "foradil/spiriva" or combined LABD and inhaled steroids "miflonide" according to GOLD recommendations peripheral muscles exercise training: (upper limb and lower limb strength and endurance training) inspiratory muscle training: (at intensity that progressively increased from 30% to 60% of patients' maximal inspiratory pressure)
  Interventions: Drug: theophylline, long acting bronchodilators (LABD) or combined LABD and inhaled steroids according to GOLD recommendations; Other: peripheral muscles exercise training; Device: inspiratory muscle training
- control positive group (group B) (Active Comparator): pharmacologic treatment: theophylline "uniphyllin", long acting bronchodilators "foradil/spiriva" or combined LABD and inhaled steroids "miflonide" according to GOLD recommendations peripheral muscles exercise training: (upper limb and lower limb strength and endurance training)
  Interventions: Drug: theophylline, long acting bronchodilators (LABD) or combined LABD and inhaled steroids according to GOLD recommendations; Other: peripheral muscles exercise training
- control negative group (group C) (Active Comparator): pharmacologic treatment: theophylline "uniphyllin", long acting bronchodilators "foradil/spiriva" or combined LABD and inhaled steroids "miflonide" according to GOLD recommendations
  Interventions: Drug: theophylline, long acting bronchodilators (LABD) or combined LABD and inhaled steroids according to GOLD recommendations

INTERVENTIONS:
Drug: theophylline, long acting bronchodilators (LABD) or combined LABD and inhaled steroids according to GOLD recommendations
  Other Names: uniphyllin, foradil, spiriva, miflonide
Other: peripheral muscles exercise training
  Arms: Study group (group A); control positive group (group B)
Device: inspiratory muscle training — Patients started breathing at a resistance that required generation of 30% of their PImax for one week. The load was then increased incrementally, 5-10%, to reach generation of 60% of their PImax at the end of the first month. Specific IMT was then continued at 60% of their PImax adjusted weekly to the new PImax achieved.
  Other Names: Threshold® Inspiratory Muscle Trainer, Healthscan, New Jersey, NJ, USA
  Arms: Study group (group A)

SUMMARY:
The aim is to study effectiveness of inspiratory muscle training as a part of exercise training in patients with Chronic Obstructive Pulmonary Disease (COPD) and if it adds to general exercise training program in regard to respiratory muscle strength, dyspnea, exercise performance and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Exsmokers
* Low PImax compared to reference values [lower limits of normal: 80 cmH2O for patients less than or equal 54 years old; 71 cmH2O for patients' age between 55-64 years; and 65 cmH2O for patients 65 years old ].
* Stable patients without history of exacerbation or hospitalization four weeks before starting the study.

Exclusion Criteria:

* Lack of motivation and compliance.
* Patients with significant reversibility following bronchodilation defined as an increase in FEV1 of more than 12% and 200 ml from the pre-bronchodilator value
* Unstable cardiac disease [severe heart failure, dangerous dysrhythmias, recent myocardial infarction or unstable angina (within 4 weeks)].
* Uncontrolled hypertension
* Recent pneumothorax (within 6 weeks)
* Recent abdominal or thoracic surgery (within 6 weeks)
* Known progressive neuromuscular disorders
* Recent gastrointestinal bleeding (within 4 weeks)
* Current smokers
* Active cancer
* Patients with advanced liver diseases, or renal impairment.
* Known connective tissue diseases
* Significant endocrinal abnormalities

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
changes in respiratory muscle strength | after 4 weeks and after 8 weeks of study
  maximal inspiratory pressure, maximal expiratory pressure
changes in perception of dyspnea | after 4 weeks and after 8 weeks of study
  modified Medical Research Council and modified Borg category scale
changes in exercise performance | after 4 weeks and after 8 weeks of study
  6-min walk test
changes in quality of life | after 4 weeks and after 8 weeks of study
  BODE index, St. George's Respiratory Questionnaire for COPD patients (SGRQ-C)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Elmorsi, MD, Study Chair — Mansoura University; Mohamad E Eldesoky, MD, Study Director — Mansoura University; Mona AA Mohsen, MD, Study Director — Mansoura University; Nesrien M Shalaby, MD, Study Director — Mansoura University; Dina A Abdallah, MSc, Principal Investigator — Mansoura University